CLINICAL TRIAL: NCT00228566
Title: A Short-term (8 Week) Open-Label Study, Followed by a Long Term Evaluation, to Assess Patient-Reported Outcomes With Armodafinil Treatment (150 to 250 mg/Day) for Excessive Sleepiness in Adults With Narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: Study to Assess Patient Reported Outcomes With Armodafinil Treatment for Excessive Sleepiness in Adults With Narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10953/3046/ES/US
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Results first posted 2010-06-25 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Excessive Daytime Sleepiness; Narcolepsy; Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS)
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy; Sleep Apnea, Obstructive | interventions — Modafinil

INTERVENTIONS:
Drug: Armodafinil

SUMMARY:
The purpose of this study is to assess patient reported outcomes with armodafinil treatment in terms of improvement in sleepiness, satisfaction with treatment, impact on ability to engage in life activities (ie, daily or work and family and/or social activities), and effects on fatigue. Clinician ratings on patient response to armodafinil treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The patient is a man or a woman aged 18 through 65 years of age (inclusive) and English-speaking.
* The patient has excessive sleepiness associated with a diagnosis of narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS) according to the International Classification of Sleep Disorders (ICSD) criteria. For OSAHS, the patient must be a regular nasal continuous positive airway pressure (nCPAP) therapy user (usage at least 4 hours/night on at least 70% of nights), must have documented adequate education and intervention efforts to encourage nCPAP therapy use, the patient's nCPAP therapy regimen must be stable for at least 4 weeks prior to study entry, and the patient's nCPAP therapy must be effective in the opinion of the investigator.
* The patient is in good health as determined by a medical and psychiatric history, clinical laboratory tests, vital signs measurements, electrocardiography (ECG), physical examination, and urine drug screen (UDS) at screening.
* If currently receiving therapy for excessive sleepiness associated with their sleep disorder, the patient is dissatisfied because of efficacy and/or safety with their current therapy (i.e., pharmacologic, nap, or bright light therapy), if taken, for excessive sleepiness associated with their sleep disorder.
* The patient has a Clinical Global Impression of Severity of Illness (CGI-S) rating at baseline of 4 or more (i.e., at least moderately ill).
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include abstinence, barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method, or intrauterine device (IUD).
* The patient must be willing and able to comply with study procedures and restrictions, including the completion of self-rating scales, and be willing to return to the study center for visits as specified in this protocol.
* The patient may have been prescribed pharmacologic therapy for excessive sleepiness associated with a sleep disorder; however, they must have undergone a washout period of at least 7 days prior to the baseline visit.

Exclusion Criteria:

Patients are excluded from participating in this study if any of the following criteria are met:

* The patient has any treated or untreated clinically significant uncontrolled medical or psychiatric conditions.
* The patient has a probable diagnosis of a current sleep disorder other than the primary diagnosis of narcolepsy, OSAHS, or other etiology for the complaint of excessive sleepiness.
* The patient consumes caffeine including coffee, tea and/or other caffeine-containing beverages or food averaging more than 600 mg of caffeine/day within 1 week of the start of study drug administration.
* The patient has a medically unexplainable positive UDS at the screening visit.
* The patient has a clinically significant deviation from normal in clinical laboratory test results, vital signs values, or physical examination findings observed at the screening visit.
* The patient has used an investigational drug within 30 days or 5 half-lives (whichever is longer) before study drug administration.
* The patient has used any prescription drugs disallowed by the protocol within 7 days before the baseline visit.
* The patient has a known or suspected hypersensitivity to armodafinil or any compound present in the study drug or related compounds.
* The patient is pregnant or lactating. (Any patients becoming pregnant during the study will be withdrawn from the study).
* The patient has any disorder (including gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
* The patient has a history of alcohol, narcotic,or any other drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM-IV) within the past 5 years.
* The patient has a history of repeated therapeutic failure to therapies for excessive sleepiness.
* The patient previously participated in a clinical study with armodafinil.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-10; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (43):
- United States (43):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Neurology Consultants of Tuscaloosa, P.C., Tuscaloosa, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - PsyPharm Clinical Research, Phoenix, Arizona
  - PsyPharm Clinical Research Inc., Tucson, Arizona
  - Neurology and Clinical Study Center, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - West Coast Clinical Trials, Inc, Long Beach, California
  - Neuro-Therapeutics, Inc, Pasadena, California
  - Penninsula Research Associates, Rolling Hills Estates, California
  - Pacific Sleep Program, San Francisco, California
  - The Sleep Disorders Center of Santa Barbara, Santa Barbara, California
  - Colorado Sleep Disorder Center, Englewood, Colorado
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Neurotrials, Inc., Atlanta, Georgia
  - Sleepmed Inc., Macon, Georgia
  - Savannah Neuurology, Savannah, Georgia
  - Evanston Northwestern Healthcare, Evanston Hospital, Evanston, Illinois
  - Convenant Clinic, Waterloo, Iowa
  - Chest Medicine Assocaites d/b/a/ Sleep Medicine Specialists, Louisville, Kentucky
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Neurocare. Inc, Newton, Massachusetts
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Neurology and Neuro Science Associates, Akron, Ohio
  - North Coast Clinical Trials, Inc., Beechwood, Ohio
  - Jonathan Schwartz, Oklahoma City, Oklahoma
  - Pacific Sleep Program, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - University Services, West Chester, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Healthstar Physicians, Morristown, Tennessee
  - Sleep Medicine of Tennesse, Nashville, Tennessee
  - Metroplex Pulmonary and Sleep Center, PA, Allen, Texas
  - FutureSearch Trials, Austin, Texas
  - Sleep Medicine Associates of Texas, P.A, Plano, Texas
  - Texas Association of Pediatric Neurology, San Antonio, Texas
  - Vermont Medical Sleep Disorders Center, Essex Junction, Vermont
  - Sleep Disorders Center of the Mid Atlantic, Vienna, Virginia
  - Pacific Institute of Medical Science, Kirkland, Washington
  - Pacific Institute of Mental Health, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 centers in the US. First participant enrolled: 5 October 2005. Last participant last visit: 27 July 2006
Pre-assignment Details: 1 female participant withdrew for noncompliance after randomization but prior to receiving study drug. The number of participants then analyzed (241) by a PGI-C rating was defined to be those participants who took at least 1 dose of study drug and had at least 1 postbaseline efficacy assessment (5 patients did not meet this requirement).
Groups:
- Armodafinil 150 to 250 mg/Day: Armodafinil 150 to 250 mg once daily in the morning
Period: Overall Study
Arm/Group | Armodafinil 150 to 250 mg/Day
Started | 247
Completed | 176
Not Completed | 71
Not completed — Adverse Event | 31
Not completed — Lack of Efficacy | 14
Not completed — Lost to Follow-up | 16
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 4
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Arm/Group | Armodafinil 150 to 250 mg/Day
Number analyzed (Participants) | 247
Age Categorical [Number; unit: participants] — 1 female participant withdrew for noncompliance after randomization but prior to receiving study drug
  participants
    <=18 years | 0
    Between 18 and 65 years | 243
    >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.53)
Gender [Number; unit: participants] — 1 female participant withdrew for noncompliance after randomization but prior to receiving study drug
  participants
    Female | 137
    Male | 109
Region of Enrollment [Number; unit: participants]
  United States | 247

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders to the Patient Global Impression of Change (PGI-C) Ratings
Description: A subjective measure (PGI-C rating) of the patient's global health, ie, a patient's rating of disease severity, as compared with a pretreatment (baseline) evaluation assessment by the patient using the Patient Global Impression of Severity of illness (PGI-S). Responders at each visit were defined as having at least minimal improvement in the severity of excessive sleepiness as compared with a pretreatment evaluation made using the PGI-S.
Time Frame: Weeks 4, 8, and 12, at 3 month intervals thereafter, and at a Final Visit (or last postbaseline observation). Evaluation continues until the Final Visit, which occurs when the product is commercially available or the marketing application is withdrawn.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 to 250 mg/Day
Number analyzed (Participants) | 241
Participants | 241
Statistical Analysis 1: Comparison: Armodafinil 150 to 250 mg/Day; This was an open label study, with all patients receiving treatment with armodafinil; Test type: Superiority or Other; Descriptive Statistics; % Responders = 201/241 = 83.4, 95% CI [78.7 to 88.1] — The Overall Endpoint includes the last postbaseline value for each patient in the full analysis set, regardless of evaluation period. The Number of Responders (at least minimal improvement) at this Overall Endpoint equaled a total of 201 patients

ADVERSE EVENTS:
Arm/Group | Armodafinil 150 to 250 mg/Day
Serious Adverse Events (participants affected / at risk) | 6/246
Other Adverse Events (participants affected / at risk) | 134/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 150 to 250 mg/Day (N=246)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Fetal growth retardation (Infections and infestations) | 1
Iliac artery occlusion (Infections and infestations) | 1
Nasal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 150 to 250 mg/Day (N=246)
Nausea (Gastrointestinal disorders) | 30
Dry mouth (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 13
Nasopharyngitis (Infections and infestations) | 35
Upper respiratory tract infection (Infections and infestations) | 21
Headache (Nervous system disorders) | 50
Dizziness (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 16
Insomnia (Psychiatric disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days